CLINICAL TRIAL: NCT04304794
Title: Prevention of Iodinated Contrast Media Induced Hyperthyroidism in Patients With Euthyroid Goiter
Brief Title: Iodinated Contrast Media Induced Hyperthyroidism
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Piotr Miskiewicz, Assistant professor, Medical University of Warsaw
Other Study IDs: ICMThyro
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hyperthyroidism/Thyrotoxicosis; Hyperthyroidism; Goiter; Iodine Induced Thyrotoxicosis; Contrast Media Adverse Reaction; Thyrotoxicosis of Other Specified Origin
Keywords: Hyperthyroidism; Iodinated contrast media; Euthyroid goiter; Thyroid nodules; Thyroid volume; Thiamazole; Sodium perchlorate
MeSH Terms: conditions — Hyperthyroidism; Thyrotoxicosis; Goiter; Euthyroid Goiter; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with prophylaxis: Group of 13 patients with euthyroid goiter who received prophylactic treatment before and after iodinated contrast medium (ICM) injection. 6 patients received thiamazole with sodium perchlorate, one day prior to ICM and for at least 14 days after for thiamazole (20-40 mg/daily) and 10 days after for sodium perchlorate (900 mg/daily). 7 patients received only thiamazole as prophylactic treatment due to lack of sodium perchlorate at the time.
  Interventions: Procedure: Administration of iodinated contrast media; Drug: Prophylactic administration of antithyroid drugs before iodinated contrast media exposure
- Group without prophylaxis: Group of 23 patients with euthyroid goiter who received no prophylactic treatment before iodinated contrast medium injection.
  Interventions: Procedure: Administration of iodinated contrast media

INTERVENTIONS:
Procedure: Administration of iodinated contrast media — Each patient was exposed on iodinated contrast medium administered during computed tomography, coronary angiography or transcatheter aortic valve implantation.
Drug: Prophylactic administration of antithyroid drugs before iodinated contrast media exposure — 13 patients received thiamazole with (6 patients) or without (7 patients) sodium perchlorate, one day prior to iodinated contrast medium (ICM) and for at least 14 days after for thiamazole (20-40 mg/daily) and 10 days after for sodium perchlorate (900 mg/daily).
  Groups: Group with prophylaxis

SUMMARY:
The proper synthesis of thyroid hormones is dependent on adequate iodine supply. The mean daily iodine intake recommended by World Health Organization is 150 mg. Iodinated contrast medium (ICM) typically contains 13 500 mg of free iodine and 15-60 g of bound iodine, an amount well above acceptable upper level. In a situation of excess iodine, thyroid discontinues the release of hormones (Wolff-Chaikoff effect), which is usually transient, although can persist causing hypothyroidism. Iodine-induced hyperthyroidism (IIH), known as the Jod-Basedow phenomenon is infrequent, but elderly patients and individuals with autonomously functioning nodular goiters are at higher risk of developing this dysfunction. According to recent studies the risk of ICM-induced hyperthyroidism appears to be low. The prevalence has not been well assessed and varies from 1 % to 10 %. Currently, there are no specific guidelines concerning the prophylactic therapy of IIH. American Thyroid Association (ATA) does not recommend routine administration of antithyroid drugs before iodinated contrast medium for all patients, however, advises to consider prophylaxis in patients at high risk of developing IIH or with cardiovascular comorbidities. ATA recommends avoidance of additional iodine and administration of b-blockers alone or with antithyroid drugs as a treatment of IIH, depending on the severity of hyperthyroidism.

This study was performed to evaluate the influence of ICM on thyroid status and advantages of prophylactic therapy during ICM exposure in patients with euthyroid goiter and cardiovascular comorbidities. The association between the incidence of IIH and thyroid volume was also assessed.

DETAILED DESCRIPTION:
Patients were divided into two subsets on the basis of received prophylactic therapy. Group with prophylaxis (13 patients) received thiamazole alone (7 patients) or with sodium perchlorate (6 patients). The prophylaxis was administered one day prior to iodinated contrast medium (ICM) and for at least 14 days after ICM for thiamazole (20-40 mg/daily) and 10 days after ICM for sodium perchlorate (900 mg/daily). Group without prophylaxis (23 patients) received no prophylactic treatment. Laboratory tests were performed before and after ICM injection in all patients from both evaluated groups. Each individual had TSH and creatinine level measured at baseline. The investigators analyzed clinical data such as age, sex, mean volume of contrast media, goiter size and patients' comorbidities. Levels of TSH, FT3 and FT4 were evaluated retrospectively at different points in time after ICM. Ultrasonography was performed in each patient to assess thyroid morphology. The investigators performed a comparison between both groups in regard to duration of overt hyperthyroidism and thiamazole treatment. Thyroid volume was compared between patients who developed hyperthyroidism after ICM injection and remained euthyroid after ICM injection. Patients diagnosed with overt hyperthyroidism were treated with thiamazole.

ELIGIBILITY:
Inclusion Criteria:

* euthyroidism at baseline (defined as TSH level within the reference range)
* diffuse or multinodular goiter
* iodinated contrast media (ICM) exposure
* time of observation after ICM exposure longer than 4 weeks

Exclusion Criteria:

* Graves' disease
* administration of thyroid hormones, glucocorticoids, iodine-containing medications or iodine contrast agent within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 36 patients (15 males) with euthyroid goiter and cardiovascular comorbidities admitted to the Institute of Cardiology between January 2015 and November 2019. The median age of treated patients was 68 years old.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Influence of iodinated contrast medium administration on thyroid function. | up to 72 weeks
  Evaluation of TSH, FT3 and FT4 levels at different points in time after iodinated contrast medium injection. Normal thyroid function was defined as TSH levels between 0.27 and 4.20 mIU/L. The reference range for fT4 and fT3 was 0.93-1.7 ng/dl and 2.0-4.4 pg/ml, respectively.
Evaluation of the association between the incidence of iodine-induced hyperthyroidism and thyroid volume. | up to 72 weeks
  Analysis of association between thyroid volume and changes in thyroid status after iodinated contrast medium injection. Normal thyroid function was defined as TSH levels between 0.27 and 4.20 mIU/L. The reference range for fT4 and fT3 was 0.93-1.7 ng/dl and 2.0-4.4 pg/ml, respectively. Subclinical hyperthyroidism was diagnosed on the basis of suppressed TSH and normal fT4 and fT3 values. Overt hyperthyroidism was defined as TSH level below lower limit and elevated fT4 and/or fT3 concentrations. Ultrasonography was performed in each patient to assess thyroid volume [ml]. Enlargement of the gland was defined as a volume exceeding 18 ml in females and 25 ml in males.
Evaluation of the association between the incidence of iodine-induced hyperthyroidism and the use of prophylactic treatment with antithyroid drugs before and after iodinated-contrast medium injection. | up to 72 weeks
  Evaluation of TSH, FT3 and FT4 levels at different points in time after iodinated contrast medium injection and comparison between groups. Normal thyroid function was defined as TSH levels between 0.27 and 4.20 mIU/L. The reference range for fT4 and fT3 was 0.93-1.7 ng/dl and 2.0-4.4 pg/ml, respectively. Subclinical hyperthyroidism was diagnosed on the basis of suppressed TSH and normal fT4 and fT3 values. Overt hyperthyroidism was defined as TSH level below lower limit and elevated fT4 and/or fT3 concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Miśkiewicz, MD, PhD, Principal Investigator — Department of Endocrinology Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: Yes
The collected data will be shared in a publication.